CLINICAL TRIAL: NCT03199391
Title: Efficacy of the BioWick SureLock Implant for the Reattachment of Soft Tissue to Bone in Subjects Undergoing Rotator Cuff Repairs
Brief Title: BioWick SureLock Clinical Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAY-001
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BioWick SureLock Implant (Experimental): All subjects are part of a single arm. All subjects received the BioWick SureLock implant.
  Interventions: Device: BioWick SureLock Implant

INTERVENTIONS:
Device: BioWick SureLock Implant — The BioWick SureLock implant is a device for shoulder and extremity surgery, constructed of Ultra High Molecular Weight Polyethylene Suture. BioWick SureLock is uniquely designed to minimize these risks by avoiding manual tensioning with an inserter mechanism that ensures that the implant is consistently deployed below the cortex.

SUMMARY:
The purpose of this study is to collect postmarket data in subjects who receive surgical treatment of a full-thickness rotator cuff tear (of at least 1.5 cm) with the BioWick™ SureLock™ implant. Both performance and safety data will be collected.

DETAILED DESCRIPTION:
Study Title Efficacy of the BioWick SureLock Implant for the Reattachment of Soft Tissue to Bone in Subjects Undergoing Rotator Cuff Repairs

Sponsor Cayenne Medical, Inc., a Zimmer Biomet company

Study Design The study is a prospective, non-randomized, open-label, single-arm study that includes both preoperative assessments and follow-up assessments at 3 months, 6 months, and 12 months.

Clinical Phase Postmarket

Number of Sites Up to ten sites in the U.S.

Study Duration per Subject Subjects will be enrolled in the study for up to 12 months.

Primary Objective The primary objective of this study is to assess survivorship (lack of reoperation/device removal) with the use of the BioWick SureLock implant.

Secondary Objective

The secondary objectives of this study are:

* To document the postmarket effectiveness of the BioWick SureLock implant using ASES scores, VR-12 scores, and VAS scores, with the corresponding assessments made at 3 months, 6 months, and 12 months postoperative.
* To document the postmarket effectiveness of the BioWick SureLock implant using range of motion (ROM) measurements with the corresponding assessments made at 3 months and 6 months postoperative.
* To document device safety via device-related adverse events reported over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of rotator cuff tear which is greater than or equal to 1.5 cm and less than or equal to 4.0 cm full thickness of either the supraspinatus or infraspinatus determined by MRI which has not been previously repaired;
2. Goutallier Stage 2 or less;
3. Patte Stage II (mid humeral head retraction);
4. Tear(s) confirmed intra-operatively by calibrated probe, tears measured in both anterior-posterior and medial-lateral planes;
5. Subject is skeletally mature at the surgical site;
6. Subject is able to read and understand the ICF and has voluntarily provided written informed consent.

Exclusion Criteria:

1. Clinical diagnosis of a rotator cuff tear of the subscapularis that requires repair (not including debridement);
2. Conditions which, in the opinion of the Principal Investigator, may limit the subject's ability or willingness to follow postoperative care or study instructions;
3. If female, subject is pregnant;
4. Presence of local or systemic infection;
5. Suprascapular nerve compression requiring release or documented by EMG-NCV;
6. Substance abuse, including tobacco, alcohol, or illicit drugs which, in the investigator's judgment, could impair healing or influence study compliance;
7. Foreign body sensitivity. If material sensitivity is suspected, testing should be completed prior to device implantation;
8. Insufficient blood supply or previous infection which may hinder the healing process;
9. Subject conditions including: insufficient quantity or quality of bone or soft tissue, or immature bone where the device may impact or disrupt the growth plate;
10. Subject is a prisoner or member of another vulnerable population;
11. Cortisone injection within 6 weeks prior to surgical treatment;
12. Use of immune suppressants or chemotherapeutic medications within the last 12 months;
13. Use of systemic corticosteroids at any daily dose for more than 1 month within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, Study Director — ryan.boylan@zimmerbiomet.com
Locations (7):
- United States (7):
  - The Orthopaedic Clinic Association, Phoenix, Arizona
  - Eisenhower Medical Center, Rancho Mirage, California
  - Orthopaedic Medical Group of Tampa Bay PA, Brandon, Florida
  - Foundation for Orthopaedic Research and Eduation, Temple Terrace, Florida
  - Norton Orthopaedics and Sports Medicine, Louisville, Kentucky
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Any screened subjects who met any of the exclusion criteria were excluded from participation in this study and were not considered enrolled subjects.
Groups:
- BioWick SureLock Implant: This arm included all subjects who were implanted with the BioWick SureLock Implant.
Period: Overall Study
Arm/Group | BioWick SureLock Implant
Started | 71
Completed | 55
Not Completed | 16
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Groups:
- BioWick SureLock Implant: This arm will include all subjects who are implanted with the BioWick SureLock Implant.
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [40.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Origin | 10
  Caucasian | 56
  Hispanic | 4
  Indian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71
Duration of Symptoms/Time Since Injury [Mean (Full Range); unit: months] | 14.9 [0.5 to 120]
Current tobacco use [Count of Participants; unit: Participants]
  No | 63
  Yes | 8
Current alcohol use [Count of Participants; unit: Participants]
  No | 33
  Yes | 38
Prior Shoulder Operations [Count of Participants; unit: Participants]
  No | 49
  Yes | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Requiring Removal or Reoperation of the Implant
Description: The primary endpoint of this study is survivorship (lack of reoperation/device removal) at 12 months postoperative. Implant survivorship for each subject was determined by whether the subject underwent a revision or reoperation of the study device. Survivorship was assessed using a Kaplan-Meier analysis. Possible scores range from 0% (lowest survivorship) to 100% (highest survivorship).
Time Frame: 12 months
Population: In the statistical analysis of the primary effectiveness endpoint of the study, only subjects with evaluable endpoint were used in the statistical analysis, i.e., a complete case analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
Participants | 69

2. Secondary Outcome: Number of Participants Not Requiring Removal or Reoperation of the Implant
Description: Implant survivorship (lack of reoperation/device removal) at 3 months and 6 months postoperative. Implant survivorship for each subject was determined by whether the subject underwent a revision or reoperation of the study device. Survivorship was assessed using a Kaplan-Meier analysis. Possible scores range from 0% (lowest survivorship) to 100% (highest survivorship).
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
Participants
  3 months | 69
  6 months | 69

3. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Patient Self-Evaluation Score
Description: Pain and function as measured by the American Society of Shoulder and Elbow Surgeons (ASES) questionnaire. ASES consists of 3 subcomponent scores including pain, instability, and activities of daily living. The pain score can be 0 to 10 with 0 being no pain and 10 being the worst pain imaginable. The instability score can be 0 to 10 with 0 being no instability and 10 being the worst instability imaginable. The activities of daily living consists of 10 questions with ordinal responses of 0, 1, 2, and 3 with 3 involving no limitation and 0 is unable to do. The 3 subcomponents combine to make the overall ASES score which can range from 0 to 100 with 0 being the worst possible score and 100 being the best.
Time Frame: Preoperative, 3 months, 6 months, 1 year
Population: The number analyzed at each interval represents the number of subjects who completed the respective follow-up visit, which may be less than the overall number of participants because of missed visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
units on a scale
  Preoperative | 44.2 (17.1)
  3 months: number analyzed (Participants) | 67
  3 months | 66.7 (19.9)
  6 months: number analyzed (Participants) | 60
  6 months | 82.9 (15.8)
  12 months: number analyzed (Participants) | 55
  12 months | 92.5 (10.2)

4. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score
Description: A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. Possible scores range from 0 (no pain) to 10 (very much pain).
Time Frame: Preoperative, 3 months, 6 months, 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
score on a scale
  Preoperative | 5.5 (2.4)
  3 months: number analyzed (Participants) | 67
  3 months | 2.1 (2.4)
  6 months: number analyzed (Participants) | 60
  6 months | 1.2 (1.6)
  1 year: number analyzed (Participants) | 55
  1 year | 0.5 (0.9)

5. Secondary Outcome: The Veterans RAND 12 (VR-12) Item Health Survey Physical Score
Description: A brief, generic, multi-use, self-administered health survey comprised of 12 items. The instruments are primarily used to measure health-related quality of life, to estimate disease burden, and to evaluate the disease-specific impact on general and selected populations. A higher VR-12 score indicates better health (0-100 scale).
Time Frame: Preoperative, 3 months, 6 months, 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
score on a scale
  Preoperative | 35.3 (8.3)
  3 months: number analyzed (Participants) | 67
  3 months | 39.9 (8.4)
  6 months: number analyzed (Participants) | 60
  6 months | 46.7 (8.7)
  1 year: number analyzed (Participants) | 55
  1 year | 49.2 (7.3)

6. Secondary Outcome: The Veterans RAND 12 (VR-12) Item Health Survey Mental Score
Description: as for outcome 5
Time Frame: Preoperative, 3 months, 6 months, 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
score on a scale
  Preoperative | 53.7 (11.3)
  3 months: number analyzed (Participants) | 67
  3 months | 54.8 (11.2)
  6 months: number analyzed (Participants) | 60
  6 months | 55.9 (9.1)
  1 year: number analyzed (Participants) | 55
  1 year | 57.0 (6.5)

7. Secondary Outcome: Range of Motion (ROM) - Active Forward Elevation
Description: Range of motion (ROM): The full movement potential of a joint, usually its range of flexion and extension. Normal range for active forward elevation is 150-180 degrees.
Time Frame: Preoperative, 3 months, 6 months, 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
degrees
  Preoperative | 116.1 (42.1)
  3 months: number analyzed (Participants) | 67
  3 months | 132.1 (30.8)
  6 months: number analyzed (Participants) | 60
  6 months | 153.4 (23.3)
  1 year: number analyzed (Participants) | 55
  1 year | 162.1 (18.7)

8. Secondary Outcome: Device Safety
Description: Safety evaluations were based on the frequency and incidence of device-related adverse events. Device-related adverse events included all reported adverse events classified as "Definitely" or "Possibly" related to the device. Adverse event data were collected throughout the entire duration of the study from enrollment thru subject completion. Routine collection occurred at each visit (3 months, 6 months, and 1 year). Additional details of reports of adverse events can be found in the Adverse Events section of the posted results.
Time Frame: 1 year
Population: All enrolled subjects were analyzed for device safety through the end of their study participation.
Measure: Number; unit: device-related adverse events
Arm/Group | BioWick SureLock Implant
Number analyzed (Participants) | 71
device-related adverse events | 8

ADVERSE EVENTS:
Time Frame: 3 months, 6 months, and 1 year
Description: Adverse event data were collected throughout the entire duration of the study from enrollment thru subject completion. Routine adverse event collection occurred at each visit (3 months, 6 months, and 1 year).
Arm/Group | BioWick SureLock Implant
All-Cause Mortality (participants affected / at risk) | 1/71
Serious Adverse Events (participants affected / at risk) | 5/71
Other Adverse Events (participants affected / at risk) | 29/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioWick SureLock Implant (N=71)
Stepped on a nail with right foot. (Infections and infestations) | 1
Increased pain, loose rotator cuff anchor (non-study device) (Musculoskeletal and connective tissue disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Chest pain and received heart catheter (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Left knee OA (Musculoskeletal and connective tissue disorders) | 1
Subject death after no longer able to breathe (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioWick SureLock Implant (N=71)
Tear and retraction of entire supraspinatus tendon (Musculoskeletal and connective tissue disorders) | 1
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 1
3 month MRI shows recurrent full-thickness tear of the supraspinatus (Musculoskeletal and connective tissue disorders) | 1
Right rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1
Worsening of left shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Patient is stiff at 3 month and 6 month visit (Musculoskeletal and connective tissue disorders) | 1
Tightness in trigger points within the cervical paraspinous muscles and levator scapular muscle (Musculoskeletal and connective tissue disorders) | 1
Right (contralateral) shoulder pain after fall (Musculoskeletal and connective tissue disorders) | 1
Neck pain - post op cervical discectomy (Nervous system disorders) | 1
Full thickness defect of the anterior supraspinatus tendon just medial to the biowick anchors (Musculoskeletal and connective tissue disorders) | 1
Left shoulder pain with certain movements (Musculoskeletal and connective tissue disorders) | 1
Patient presented with ipsilateral bursitis/adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 1
Headaches for 2 weeks (General disorders) | 1
Patient healed quickly and subsequently developed capsulitis (Musculoskeletal and connective tissue disorders) | 1
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Medial meniscus tear on right knee (Musculoskeletal and connective tissue disorders) | 1
Patient fell off bike and ruptured his achilles tendon (Musculoskeletal and connective tissue disorders) | 1
Metal shaving in left 3rd toe (General disorders) | 1
Increased pain in right shoulder and neck radiating to fingers (Musculoskeletal and connective tissue disorders) | 1
Presented to the ed with complaints of cough and wheezing x 2 weeks (Respiratory, thoracic and mediastinal disorders) | 1
At 3 month visit, patient is noted to be stiff (Musculoskeletal and connective tissue disorders) | 1
Melanoma excision on right shoulder (Skin and subcutaneous tissue disorders) | 1
Patient developed lateral epicondylitis of right humerus (Musculoskeletal and connective tissue disorders) | 1
6 month MRI report notes a re-tear of the supraspinatus and associated bursal-sided fluid build-up (Musculoskeletal and connective tissue disorders) | 1
Sharp stabbing pain down middle of back. Preexisting back pain got much worse right after surgery (Nervous system disorders) | 1
Adhesive capsulitis/arthro fibrosis diagnosed. (Musculoskeletal and connective tissue disorders) | 1
Loosened posterior superior anchor with fluid collection and retraction. (Musculoskeletal and connective tissue disorders) | 1
Worsening of lumbar degenerative disc disease (Nervous system disorders) | 1
Capsulitis/stiffness. Required cortisone injection (Musculoskeletal and connective tissue disorders) | 1
3/4 weeks post-op, patient developed erythema. Required surgical debridement and ROH. (Musculoskeletal and connective tissue disorders) | 1
Patient presented to the pain clinic with known history of migraine headaches (Musculoskeletal and connective tissue disorders) | 1
New full-thickness tear at the supraspinatus/infraspinatus junction from shoveling. (Musculoskeletal and connective tissue disorders) | 1
Low back pain with radiation into left thigh (Nervous system disorders) | 1
Neck pain and decreased ROM related to degenerative cervical disc disease (Nervous system disorders) | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1
3 month MRI reports recurrent tear which becomes symptomatic sometimes (Musculoskeletal and connective tissue disorders) | 1
R shoulder pain/difficulty with throwing activities and shoulder movement (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
New tenderness of left shoulder (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT03199391/Prot_SAP_000.pdf